CLINICAL TRIAL: NCT07173985
Title: Strategies for Optimizing a Mailed FIT Program in Appalachia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul Reiter, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: OSU-24377; R01CA282162 (NIH)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not aware of the research questions being tested in the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (standard FIT kit plus telephone PN) (Experimental): Participants receive standard FIT kit plus telephone patient navigation (PN)
  Interventions: Behavioral: Standard FIT kit; Behavioral: Telephone patient navigation
- Group B (standard FIT kit plus text message PN) (Experimental): Participants receive standard FIT kit plus text message patient navigation (PN)
  Interventions: Behavioral: Standard FIT kit; Behavioral: Text message patient navigation
- Group C (enhanced FIT kit plus telephone PN) (Experimental): Participants receive enhanced FIT kit plus telephone patient navigation (PN)
  Interventions: Behavioral: Enhanced FIT kit; Behavioral: Telephone patient navigation
- Group D (enhanced FIT kit plus text message PN) (Experimental): Participants receive enhanced FIT kit plus text message patient navigation (PN)
  Interventions: Behavioral: Enhanced FIT kit; Behavioral: Text message patient navigation

INTERVENTIONS:
Behavioral: Standard FIT kit — Receive a standard FIT kit
  Arms: Group A (standard FIT kit plus telephone PN); Group B (standard FIT kit plus text message PN)
Behavioral: Enhanced FIT kit — Receive a enhanced FIT kit that includes a video brochure, disposable gloves, and a disposable stool collection device
  Arms: Group C (enhanced FIT kit plus telephone PN); Group D (enhanced FIT kit plus text message PN)
Behavioral: Telephone patient navigation — Receive telephone-based patient navigation
  Arms: Group A (standard FIT kit plus telephone PN); Group C (enhanced FIT kit plus telephone PN)
Behavioral: Text message patient navigation — Receive text message-based patient navigation
  Arms: Group B (standard FIT kit plus text message PN); Group D (enhanced FIT kit plus text message PN)

SUMMARY:
The proposed study is examining strategies for optimizing mailed fecal immunochemical test (FIT) programs. In doing so, it will assess the efficacy of two promising strategies, FIT kit materials and patient navigation delivery mode. These strategies may help to improve colorectal cancer screening rates.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Determine the efficacy of two strategies for increasing colorectal cancer screening.

OUTLINE: Participants are randomized to 1 of 4 groups.

GROUP I: Participants receive a standard FIT kit plus telephone patient navigation.

GROUP II: Participants receive a standard FIT kit plus text message patient navigation.

GROUP III: Participants receive an enhanced FIT kit plus telephone patient navigation.

GROUP IV: Participants receive an enhanced FIT kit plus text message patient navigation.

ELIGIBILITY:
Inclusion Criteria:

* Resident of an Appalachian county
* Medical visit at a participating health system in the past two years
* Average-risk for colorectal cancer
* Not currently within colorectal cancer screening guidelines

Exclusion Criteria:

-

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
FIT Return | Within 8 weeks of FIT kit distribution
  Proportion of participants who return of a completed FIT kit

CONTACTS AND LOCATIONS:
Overall Officials: Paul Reiter, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu